CLINICAL TRIAL: NCT00637650
Title: Should we Strive for Absolute "Stone Freedom" While Performing Holmium Laser Lithotripsy for Ureteral Stones? A Randomized Controlled Trial.
Brief Title: Management of Fragments During Ureteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Chaim Sheba Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 4638
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Urinary Stones
MeSH Terms: conditions — Urinary Calculi | interventions — Ureteroscopy

ARMS (2):
- B (Experimental): Experimental group: patients in whom "stone dust" was left for spontaneous elimination
  Interventions: Procedure: Ureteroscopy, Holmium laser lithotripsy, no intent to retrieve any remaining fragment
- A (Other): Control group: Patients in whom all fragments resulting from laser lithotripsy of ureteral stones were actively retrieved
  Interventions: Procedure: Ureteroscopy, Holmium Laser lithotripsy and active retrieval of fragments

INTERVENTIONS:
Procedure: Ureteroscopy, Holmium Laser lithotripsy and active retrieval of fragments
  Arms: A
Procedure: Ureteroscopy, Holmium laser lithotripsy, no intent to retrieve any remaining fragment
  Arms: B

SUMMARY:
The purpose of this study is to study the outcome of patients after ureteroscopy in which all fragments remaining after holmium laser lithotripsy were retrieved compared to those where small, insignificant fragments were left for spontaneous passage.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ureteral stones suitable for endoscopic treatment

Exclusion Criteria:

* presence of ipsilateral kidney stones
* known ureteral stricture
* previous placement of ureteral stent
* use of drugs with known activity on smooth ureteral muscle
* unwillingness or impossibility to return for follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
unplanned medical visits | 30 days

SECONDARY OUTCOMES:
Hospital Admissions, need for pain killers, time to complete recovery | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Chaim Sheba Medical Center, Tel Litwinsky, Ramat Gan, Israel